CLINICAL TRIAL: NCT01639677
Title: Randomized Clinical Trial Between Laparoscopic Gastric Bypass and Laparoscopic Vertical Banded Gastroplasty for Morbid Obesity
Brief Title: Clinical Trial Between Laparoscopic Gastric Bypass and Laparoscopic Vertical Banded Gastroplasty for Morbid Obesity
Acronym: LOK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Torsten Olbers, MD, PhD, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOK-2
Record Dates: First submitted 2011-09-22; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Morbid Obesity
Keywords: Obesity; weight loss; surgery; gastric bypass; VBG
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic gastric bypass (Experimental)
  Interventions: Procedure: Laparoscopic gastric bypass
- Laparoscopic VBG (Active Comparator): Laparoscopic vertical banded gastroplasty
  Interventions: Procedure: Laparoscopic VBG

INTERVENTIONS:
Procedure: Laparoscopic gastric bypass — Laparoscopic gastric bypass surgery
  Arms: Laparoscopic gastric bypass
Procedure: Laparoscopic VBG — Laparoscopic vertical banded gastroplasty
  Arms: Laparoscopic VBG

SUMMARY:
This is a randomized clinical trial assessing the outcome of two surgical strategies to treat severe obesity; laparoscopic gastric bypass and laparoscopic VBG. Main outcome is weight loss and weight loss maintenance but other factors as body composition, eating pattern, metabolic normalisation, energy expenditure will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-50 kg/m2
* 20-60 y

Exclusion Criteria:

* Severe co-morbidity
* Unmotivated to long term follow up

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2000-04; Primary Completion 2001-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1, 2, 5 and 10 years after surgery

SECONDARY OUTCOMES:
Body composition | 1, 2, 5 and 10 years after surgery
Eating pattern | 1, 2, 5 and 10 years after surgery
Energy expenditure | 1, 2, 5 and 10 years after surgery
Gut hormonal response | 4 and 10 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Olbers, MD, PhD, Principal Investigator — GöteborgU
Locations (1):
- Department of Surgery, Gothenburg, Gothenburg, Sweden